CLINICAL TRIAL: NCT04055545
Title: 12 Week High Intensity Interval Training VS Moderate Intensity Continuous Training in Chronic Low Back Pain Subjects: a Randomized Single-blinded Feasibility Study
Brief Title: High Intensity Interval Training VS Moderate Intensity Continuous Training in Chronic Low Back Pain Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cerini Tamara (Other)
Collaborators: Schulthess Klinik (Other)
Responsible Party: Sponsor-Investigator, Cerini Tamara, Sponsor-Investigator, HES-SO Valais-Wallis
Organization: HES-SO Valais-Wallis (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HIITvsMICT
Record Dates: First submitted 2019-08-10; First posted 2019-08-13 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MICT (Active Comparator)
  Interventions: Other: MICT
- HIIT (Active Comparator)
  Interventions: Other: HIIT

INTERVENTIONS:
Other: HIIT — * 5 min. warm up
  * 10 × 60 seconds burst
  * 60 seconds recovery after each burst
  * Burst phase: HRR >90%
  * Recovery phase: HRR btw. 30-39%
  * 5 min. cool down
  Other Names: high intensity interval training
  Arms: HIIT
Other: MICT — * 5 min. warm up
  * 20 min. continuous cycling: HRR btw. 40% - 59%
  * 5 min. cool down
  Other Names: moderate intensiv continuous training
  Arms: MICT

SUMMARY:
The current guidelines for non-specific CLBP, recommend a conservative approach with exercise therapy, as first line treatment. Endurance and resistance training are two examples of recommended exercise therapies. However, it appears that none is recommended as superior over the other.

DETAILED DESCRIPTION:
The lack of studies using HIIT in CLBP subjects, is the reason why it is needed to conduct an investigation about its effects.

However, firstly it is needed to assess the feasibility and safety of the HIIT protocol, to integrate it in the daily practise and future research.

In a single-center, single-blinded randomized feasiblity study, the investigators aim to prove the feasibility and safety of a 12 week HIIT programm.

ELIGIBILITY:
Inclusion Criteria:

* Oswestry disability index (ODI) Score ≥ 14%
* Low back pain for at least 3 months.
* Declared suitable by their physician or hospital consultant to start an exercise programme and to perform a graded exercise testing to determine the heart rate peak.
* Good understanding of German or English, written and spoken.
* Age between 29 - 69
* No or stopped physical therapy.

Exclusion Criteria:

* Pre-existing unstable heart disease or suspected angina pectoris, cardiac dysrhythmias, heart failure, aneurysm or aortic stenosis.
* Known pregnancy.
* Previous low back spinal surgery in the last 2 years.
* Tumour, spinal stenosis, spinal fractures or radiculopathy.
* Comorbid health conditions like diabetes mellitus, rheumatoid arthritis or other systemic inflammatory diseases.

Ages: 29 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Adherence | 13 weeks
  Difference in training adherence rate between HIIT and MICT. The adherence rate will be calculated in the amount of days a patient trained versus the total days they were scheduled to train.

SECONDARY OUTCOMES:
Enjoyability | 13 week
  Likert scale from -3 to +3. -3 = I hate it, 0 = Neutral, +3 = I enjoy it.
Willingness to continue the training | 13 weeks
  Likert scale from -3 to +3. -3 = Very low, 0 = Neutral, +3 = Very high.
Number of Adverse Events & Dropout rate | 13 weeks
  Dropout rate and adverse events connected with the training
Recruited rate | 3 months
  Screened patients in relation with the number of recruited patients

OTHER OUTCOMES:
Oswestry disability index | 13 weeks
  The Oswestry low back pain disability questionnaire examines the perceived level of disability in the everyday activities of daily living. 0% to 20% = Minimal disability; 21% to 40% = Moderate disability; 41% to 60% = Severe disability; 61% to 80% = crippled; 81% to 100%.
Numeric Pain Rate Scale | 13 weeks
  Pain score from 0 to 10. 0 = No pain, 5 = Moderate pain, 10 = Worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cerini T, Hilfiker R, Riegler TF, Felsch QTM. 12 weeks high intensity interval training versus moderate intensity continuous training in chronic low back pain subjects: a randomised single-blinded feasibility study. Arch Physiother. 2022 May 2;12(1):12. doi: 10.1186/s40945-022-00136-3. PMID 35491417